CLINICAL TRIAL: NCT05128435
Title: Coronavirus Pediatric Serological Study
Acronym: CoPSS
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire Saint Pierre (Other)
Responsible Party: Principal Investigator, Lisa Tomasi, Doctor (pediatrician), Centre Hospitalier Universitaire Saint Pierre
Other Study IDs: 200629
Record Dates: First submitted 2021-10-28; First posted 2021-11-22 (Actual); Last update posted 2021-11-22 (Actual); Status verified 2021-11

CONDITIONS: SARS-CoV2 Infection
Keywords: SARS-CoV-2; Immune response; Children
MeSH Terms: conditions — COVID-19 | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Positive Children: Children under 15 years old tested positive for SARS-CoV-2 by PCR on nasopharyngeal swab
  Interventions: Diagnostic Test: Blood sample

INTERVENTIONS:
Diagnostic Test: Blood sample — Blood sample taken 3 to 5 months after the infection

SUMMARY:
The Coronavirus Pediatric Serological Study's aim is to provide a better insight of children's immune response after SARS-CoV-2 infection.

Serological tests were conducted on blood samples taken 3 to 5 months after the children's viral infection.

The study was performed in collaboration with the Institute of Medical Immunology, were antibody levels were measured and immunoglobulin subclasses profiles were studied.

DETAILED DESCRIPTION:
The hospital laboratory provided us the list of children under 15 years old tested for SARS-CoV-2 in Saint-Pierre Hospital (Brussels) by PCR on nasopharyngeal swab between March 1 2020 and December 31 2020.

The medical files of all children that were tested positive for SARS-CoV-2 were reviewed and clinical information was collected.

For each positive child, the family was contacted by phone 3 months after the proven viral infection in order to ask permission to take a single blood test.

Covid19 serologies were performed in the hospital laboratory, and blood samples were then sent to the Institute of Medical Immunology, were antibody levels and immunoglobulin subclasses were studied.

ELIGIBILITY:
Inclusion Criteria:

- Tested positive for SARS-CoV-2 by PCR on naso-pharyngeal swab performed in Saint-Pierre Hospital (Brussels) between March 1 2020 and December 31 2020

Exclusion Criteria:

* /

Ages: 0 Months to 179 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children under 15 years old
Sampling Method: Non-Probability Sample
Enrollment: 49 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2021-05-31 (Actual)

PRIMARY OUTCOMES:
SARS-CoV-2 antibody levels in asymptomatic patients | 3 to 5 months after SARS-CoV-2 infection
  Measurement of SARS-CoV-2 IgG (total and subclasses), IgA (total and subclasses) and IgM levels in the sera of children who did not show any symptoms at the time of the viral infection
SARS-CoV-2 antibody levels in mildly symptomatic patients | 3 to 5 months after SARS-CoV-2 infection
  Measurement of SARS-CoV-2 IgG (total and subclasses), IgA (total and subclasses) and IgM levels in the sera of children presenting mild symptoms at the time of the viral infection
SARS-CoV-2 antibody levels in hospitalized patients | 3 to 5 months after SARS-CoV-2 infection
  Measurement of SARS-CoV-2 IgG (total and subclasses), IgA (total and subclasses) and IgM levels in the sera of children who required an hospitalisation at the time of the viral infection

CONTACTS AND LOCATIONS:
Locations (1):
- Saint-Pierre Hospital, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: Undecided